CLINICAL TRIAL: NCT00719277
Title: Pilot Clinical Study of the Sleuth Implantable ECG Monitoring System
Brief Title: Feasibility Study: Sleuth Monitoring System
Acronym: PULSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Transoma Medical (Industry)
Responsible Party: Wim Stegink, Transoma Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP-005
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Arrhythmia; Syncope
Keywords: cardiac arrhythmia; syncope; ECG; implantable ECG monitor; ILR
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sleuth Implantable ECG Monitoring System — The study device provides monitoring only. It cannot provide intervention or treatment.

SUMMARY:
The purpose of the study is to evaluate the safety and performance of the Sleuth Monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18 years at time of enrollment
* Either of the following:

  1. MI > 30 days prior to enrolment and LVEF < = 35% by echocardiography (or nuclear imaging as necessary)
  2. Syncope of unknown etiology

Exclusion Criteria:

* Life expectancy < 12 months following enrollment
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-07 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostically viable ECG signals | daily

SECONDARY OUTCOMES:
rate of device-related adverse events | 1, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wim Stegink, Study Director — Transoma Medical
Locations (1):
- Hospital Paitilla, Panama City, Panama